CLINICAL TRIAL: NCT07016776
Title: Evaluation of the Association Between Uroflowmetry Curve Patterns and IPSS Domains in Men With Lower Urinary Tract Symptoms
Brief Title: Uroflowmetry Curve Types and IPSS in Men With LUTS
Acronym: UROFLOW-IPSS
Status: Not yet recruiting | Type: Observational
Sponsor: Tarik Emre Sener (Other)
Responsible Party: Sponsor-Investigator, Tarik Emre Sener, Assoc. Prof., Marmara University
Organization: Marmara University (Other)
Other Study IDs: MAR.UAD.0022
Record Dates: First submitted 2025-05-30; First posted 2025-06-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lower Urinary Tract Symptoms (LUTS); Benign Prostatic Hyperplasia (BPH); Voiding Dysfunction
Keywords: International Prostate Symptom Score (IPSS); Uroflowmetry; Flow curve pattern; Male urinary symptoms; Prospective observational study
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with LUTS (Lower Urinary Tract Symptoms): Male patients aged 40 years and older presenting with lower urinary tract symptoms (LUTS), evaluated using the International Prostate Symptom Score (IPSS), uroflowmetry, and standard clinical parameters. All participants will be classified based on their uroflowmetry curve type and IPSS subdomain scores (storage and voiding symptoms).

SUMMARY:
This prospective observational study aims to evaluate the relationship between different uroflowmetry curve types and International Prostate Symptom Score (IPSS) domains in men presenting with lower urinary tract symptoms (LUTS). Participants will undergo routine clinical evaluations including uroflowmetry, laboratory assessments, and completion of the IPSS questionnaire.

Each participant will be classified into one of five predefined uroflowmetry curve types (normal/bell-shaped, plateau, staccato, intermittent, or tower-like). The IPSS will be analyzed both as a total score and as two subdomains: storage and voiding symptoms. Additional data such as age, comorbidities, medication use, prostate volume, eGFR, and QoL score will also be recorded to assess potential correlations and predictive factors for symptom severity.

The goal of this study is to better understand how objective urodynamic findings correlate with patient-reported symptoms and to inform clinical decision-making in men with LUTS.

DETAILED DESCRIPTION:
This is a single-center, prospective, cross-sectional observational study conducted at Marmara University, Faculty of Medicine, Department of Urology. The study includes male patients aged 40 years and older presenting with lower urinary tract symptoms (LUTS) who are capable of completing the International Prostate Symptom Score (IPSS) questionnaire and undergoing uroflowmetry.

The primary objective is to evaluate the association between uroflowmetry curve types and IPSS scores, particularly focusing on the IPSS storage domain (questions 2, 4, 7), voiding domain (questions 1, 3, 5, 6), and the total score. Patients will be classified according to five uroflowmetry curve patterns: 1) normal (bell-shaped), 2) plateau, 3) staccato, 4) interrupted/intermittent, and 5) tower-like.

Demographic and clinical data will be collected including age, height, weight, smoking status, comorbidities (HTN, DM, CHF/CAD), history of urinary tract infections or retention, medication use (alpha-blockers, 5-ARI, anticholinergics), and medication adherence. Objective parameters such as prostate volume, PSA, serum creatinine, and estimated glomerular filtration rate (eGFR) will also be recorded.

The study will explore statistical associations between uroflowmetry curve types and symptom severity across the IPSS domains. The goal is to identify specific curve types that may correlate with increased symptom burden and/or predict surgical preference. Data analysis will include descriptive statistics, correlation analysis, and regression modeling as appropriate.

This study does not involve any experimental intervention and poses minimal risk to participants. All procedures and assessments are part of routine clinical practice. Ethical approval has been obtained, and informed consent will be acquired from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Male patients aged 40 years or older
* Presenting with lower urinary tract symptoms (LUTS)
* Able to complete the IPSS questionnaire
* Underwent uroflowmetry and serum creatinine testing

Exclusion Criteria:

* History of prior prostate surgery
* Active urinary tract infection
* Known diagnosis of neurogenic bladder
* Current use of indwelling urinary catheter

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male outpatients aged 40 years and older with LUTS who presented to the urology department of a tertiary academic center.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Association between uroflowmetry curve type and total IPSS score | At baseline (single time point)
  Assessment of the relationship between different uroflowmetry curve patterns (normal, plateau, staccato, intermittent, tower) and total International Prostate Symptom Score (IPSS) in men with LUTS.

SECONDARY OUTCOMES:
Association between uroflowmetry curve type and IPSS storage symptom sub-score | At baseline
  Evaluation of the correlation between flow curve pattern and IPSS storage domain (questions 2, 4, and 7).
Association between uroflowmetry curve type and IPSS voiding symptom sub-score | At baseline
  Evaluation of the correlation between flow curve pattern and IPSS voiding domain (questions 1, 3, 5, and 6).

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to the lack of a formal data sharing platform. However, de-identified data may be provided upon reasonable request by qualified researchers, in line with ethical approval and institutional policies.

REFERENCES:
- [Result] Tarcan, T., et al. (2024). "ICS educational module: The practice of uroflowmetry in adults." Continence 9: 101065

DOCUMENTS (1):
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT07016776/ICF_000.pdf